CLINICAL TRIAL: NCT05426941
Title: Feasibility and Acceptability of Music Imagery, and Listening Interventions for Analgesia (FAMILIA)
Brief Title: Feasibility and Acceptability of Music Therapy for Chronic Pain
Acronym: FAMILIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); Indiana Institute for Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1863501-22-C-20
Record Dates: First submitted 2022-05-25; First posted 2022-06-22 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music Imagery (Experimental): MI sessions will be delivered by board-certified music therapists with specialized training in MI and the study treatment protocol.The 8-session protocol has two stages. Stage 1 (sessions 1-4) is focused on learning to use music and imagery for self-regulation. Once the Veteran has demonstrated skill in using music for self-regulation, Stage 2 (sessions 5-8) shifts to identify and deepen their inner resources and how they can use those resources for self-care.
  Interventions: Behavioral: Music Imagery
- Music Listening (Experimental): Following a one-time meeting with a music therapist, an electronic playlist will be compiled for the Veteran to listen to during the 12-week treatment period.
  Interventions: Behavioral: Music Listening
- Usual care (No Intervention): Participants in the usual care arm (as is the case for MI and ML groups) may receive analgesics and non-pharmacological treatments (e.g., physical therapy) for their chronic musculoskeletal pain.

INTERVENTIONS:
Behavioral: Music Imagery — Up to 30 participants will be randomized to receive 8 weekly Music Imagery sessions over 8-12 weeks.
  Other Names: music therapy
  Arms: Music Imagery
Behavioral: Music Listening — Up to 15 participants will be randomized to independent music listening.
  Other Names: music therapy
  Arms: Music Listening

SUMMARY:
The purpose of the study is to examine the feasibility and acceptability of two music interventions delivered through telehealth for chronic musculoskeletal pain. This pilot study evaluates outcomes (feasibility, acceptability, pain and associated outcomes) in a single-component, minimally interactive music listening (ML) intervention and a multi-component, more interactive music imagery (MI) intervention.

DETAILED DESCRIPTION:
FAMILIA is a 3-arm, parallel group, pilot trial. Sixty Veterans will be randomized to one of three conditions: MI, ML, or usual care. Aim 1 is to test the feasibility and acceptability of a multi-component, interactive MI intervention (8-weekly, individual sessions) and a single-component, minimally interactive ML intervention (independent music listening). Feasibility metrics related to recruitment, retention, engagement, and completion of treatment protocol and questionnaires will be assessed. Up to 20 qualitative interviews will be conducted to assess Veteran experiences with both interventions, including perceived benefits, acceptability, barriers, and facilitators. Interview transcripts will be coded and analyzed for emergent themes. Aim 2 is to explore the effects of MI and ML versus usual care on pain and associated patient-centered outcomes. These outcomes and potential mediators will be explored through changes from baseline to follow-up assessments at 1, 3, and 4 months. Descriptive statistics will be used to describe outcomes; this pilot study is not powered to detect differences in outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (> 6 months) musculoskeletal pain of at least moderate severity (≥5 on 0-10 numeric scale)
* Access to a personal computer, tablet computer, and/or smartphone,
* Ability to pass technology assessment screen, and
* Not currently receiving music therapy services

Exclusion Criteria:

* Serious or unstable medical (e.g., Congestive Heart Failure, Chronic Obstructive Pulmonary Disease) or psychiatric illness (e.g., psychosis, mania) or housing insecurity that could compromise study participation,
* Suicidal ideation with current intent/plan,
* Hearing or cognitive impairment that may interfere with music listening or abstract thinking needed for imagery work,
* Lack access to a personal computer, tablet computer, and/or smartphone,
* Unable to pass technology assessment screen, or
* Currently receiving music therapy services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of contacted and eligible Veterans consent to study participation, attend intervention sessions, and complete the treatment protocol and scheduled outcome assessments? | at 3 months
  Determine the feasibility of the music therapy interventions
Aspects of the interventions do Veterans perceive to be most/least helpful or most/least liked? | at 3 months
  Assess participant acceptability of the music therapy interventions

SECONDARY OUTCOMES:
Numeric Rating Scale for Pain intensity | Baseline, 1, 3, and 4 months
  assessment of severity of pain, scored 0 to 10 with higher scores representing more intense pain
Brief Pain Inventory - Pain interference subscale | Baseline, 1, 3, and 4 months
  how does pain interfere with 7 activities, scored 0 to 10 with higher scores representing more interference of pain with activities
Brief Pain Catastrophizing Scale | Baseline, 1, 3, and 4 months
  assessment of pain belief, scored 0 to 12 with higher scores representing more pain catastrophizing (worse outcome)
Centrality of Pain Scale | Baseline, 1, 3, and 4 months
  assessment of pain coping, scored 10 to 50 with higher scores representing the belief that pain is central to individual's life (worse outcome)
Patient Global Impression of Change Scale | 1,3 and 4 months
  assessment of treatment response, scored 1 to 7 with higher scores representing greater improvement from starting the intervention
PROMIS Sleep Scale | Baseline, 1, 3, and 4 months
  assessment of sleep quality, scored 1 to 5 with higher scores representing worse sleep quality (worse outcome)
PHQ-9 Depression Measure | Baseline, 1, 3, and 4 months
  assessment of depression severity, scored 0 to 27 with higher scores representing more severe depression (worse outcome)
GAD-7 Anxiety Measure | Baseline, 1, 3, and 4 months
  assessment of anxiety severity, scored 0 to 21 with higher scores representing more severe anxiety (worse outcome)
Perceived Stress Scale | Baseline and 3 months
  assessment of stress severity, scored 0 to 14 with higher scores representing more severe stress (worse outcome)
EQ 5D Scale for Health-Related Quality of Life | Baseline and 3 months
  assessment of generic health-related quality of life, higher scores represent improved quality of life
EQ 5D Scale for Health-Related Quality of Life | Baseline and 3 months
  assessment of generic health-related quality of life, scored 0 to 100 with higher scores represent improved quality of life (better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Bair, Principal Investigator — Roudebush VA Medical Center; Maya Story, Principal Investigator — Roudebush VA Medical Center
Locations (1):
- Roudebush VA Medical Center, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Story KM, Wasmuth S, Belkiewitz JM, Whalen C, Robb SL, Bravata DM, Bair MJ. Military veterans' perspectives on using music to manage chronic pain: themes from the feasibility and acceptability of music imagery and listening interventions for analgesia study. Front Neurol. 2025 Aug 6;16:1613220. doi: 10.3389/fneur.2025.1613220. eCollection 2025. PMID 40843263
- [Derived] Story KM, Bravata DM, Robb SL, Wasmuth S, Slaven JE, Whitmire L, Barker B, Menen T, Bair MJ. Feasibility and Acceptability of Music Imagery and Listening Interventions for Analgesia: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Sep 22;11(9):e38788. doi: 10.2196/38788. PMID 36136377